CLINICAL TRIAL: NCT01878981
Title: Health Economics Evaluation of Catheter Ablation Versus Drug Therapy in Atrial Fibrillation (AF) in China
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: CAAF 2011
Record Dates: First submitted 2013-05-29; First posted 2013-06-17 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation versus Drug Therapy in AF in China
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To generate real world evidence to compare clinical outcomes and patient health-related quality of life, resulting from catheter ablation therapy with clinical outcome and patient health-related quality of life resulting from drug therapy in China. An economic model will be constructed, and using the clinical events evidence collected in this study, and China long-term disease progression and local disease cost data to perform a cost-effectiveness evaluation of Catheter Ablation versus Drug Therapy in AF (Paroxysmal plus Persistent AF) patients.

DETAILED DESCRIPTION:
The evidence generated by this study is expected to help inform medical decision makers with the clinical and economic data of therapy for AF patients, and also provide policy decision makers with information that can be considered /used to allocate funds for AF ablation and permit patients to have access to appropriate treatment options for AF management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent AF eligible for catheter ablation
* Age 18 to 80 years
* Able and willing to comply with all pre,post and follow-up testing and requirements.
* Be able to sign IRB/EC approved informed consent form.

Exclusion Criteria:

* Terminal illness with a life expectancy less than 1 year.
* New York Heart Association (NYHA) Class III or IV
* Previous recipient of catheter ablation therapy for AF
* Bradycardia and previous recipient of pacemaker therapy
* Previous recipient RFCA or ICD therapy
* Uncontrolled hypertension
* Recent cardiac events including MI, PCI, or valve or bypass surgery in the preceding 3 months
* Patients with serious hepatic and renal diseases
* Pregnant or prepare to be pregnant in one year
* For drug therapy arm, if the subject cannot be contacted via phone or the subject shows his/her disagreement to this study at 30 day window, the subject will be withdrawn from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 300 subjects in the catheter ablation arm (150 paroxysmal AF patients and 150 persistent AF patients) and 150 subjects in the drug treatment arm (75 paroxysmal AF patients and 75 persistent AF patients).
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2013-11-23 (Actual); Study Completion 2013-11-23 (Actual)

PRIMARY OUTCOMES:
the frequency of recurrence | 9 months followup after baseline
  the frequency of recurrence of Atrial Fibrillation/Flutter/Tachycardia

SECONDARY OUTCOMES:
Rate | 9 month follow up after baseline
  Total mortality
total cost | 9 months follow up
  Average total costs of ablation vs. drug therapy per patient
Rate | 9 months follow up from baseline
  Stroke
Rate | 9 months from baseline
  Cardiovascular death/Arrhythmic death or Cardiac arrest/Heart failure death
Duration | 9 months from baseline
  Cardiovascular or Cerebrovascular hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, doctor, Principal Investigator — Beijing Anzhen Hospital

REFERENCES:
- [Derived] Du X, Guo L, He X, Jia Y, Wu J, Long D, Yu R, Sang C, Liu X, Yin H, Xuan J, Dong J, Ma C. A comparison of the real world effectiveness of catheter ablation and drug therapy in atrial fibrillation patients in a Chinese setting. BMC Cardiovasc Disord. 2017 Jul 27;17(1):204. doi: 10.1186/s12872-017-0634-y. PMID 28750608